CLINICAL TRIAL: NCT04421508
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Pulsed, Inhaled Nitric Oxide (iNO) Versus Placebo in Subjects With Mild or Moderate Coronavirus (COVID-19)
Brief Title: A Study to Assess Pulsed Inhaled Nitric Oxide vs Placebo in Subjects With Mild or Moderate COVID-19
Acronym: COViNOX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Bellerophon Pulse Technologies (Industry)
Responsible Party: Sponsor
Organization: Bellerophon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PULSE-CVD19-001
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Coronavirus; Coronavirus Infection
Keywords: COVID; Sars-CoV-2; iNO; INOpulse; Severe Acute Respiratory Syndrome (SARS) Pneumonia; Severe Acute Respiratory Syndrome Coronavirus 2; SARS-CoV 2; COViNOX; pulsed inhaled nitric oxide; inhaled nitric oxide; portable pulsed inhaled nitric oxide; nitric oxide
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome; Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inhaled Nitric Oxide (iNO) (Active Comparator): Pulsed inhaled iNO 125 mcg/kg IBW/hour
  Interventions: Combination Product: INOpulse
- Placebo (Sham Comparator): Pulsed inhaled N2, 99.999% gas
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: INOpulse — Subjects will be treated by means of an INOpulse device using an INOpulse nasal cannula.
  Arms: Inhaled Nitric Oxide (iNO)
Combination Product: Placebo — Subjects will be treated by means of an INOpulse device using an INOpulse nasal cannula.
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled study to assess the efficacy and safety of pulsed inhaled iNO compared to placebo in subjects with COVID-19.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to assess the efficacy and safety of pulsed iNO compared to placebo in subjects with COVID-19 who are hospitalized and require supplemental oxygen without assisted ventilation. Subjects will be randomized to receive placebo or iNO125 mcg/kg ideal body weight (IBW)/hour 24 hours daily up to 14 days or until resolution or discharge.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* At least 18 years old
* Subjects must be hospitalized and have the following:

  * proven or high suspicion of SARS-CoV-2 infection and,
  * requiring oxygen supplementation defined as:
  * SpO2 ≤ 92% regardless of supplemental oxygen (ie on room air or on oxygen), or
  * SpO2 ≥ 92% on supplemental O2 and in the opinion of the Investigator it is not safe to decrease or remove the supplemental oxygen
  * require supplemental oxygen of no more than 10 L/minute, and
  * radiologic suspected or proven COVID-19 pneumonitis (chest x-ray or CT scan)
* Female subjects must have a negative pregnancy test
* Willing and able to comply with the treatment schedule and study procedures

Exclusion Criteria:

* Participating in another clinical trial of an investigational treatment for COVID-19
* Methemoglobin > 3%
* Evidence of severe multi organ failure
* Use of assisted ventilation prior to initiation of iNO
* Pregnancy or positive pregnancy test pre-dose
* Open tracheostomy
* Chronic use of a nitric oxide donor agent such as nitroglycerin or drugs known to increase methemoglobin such as lidocaine, prilocaine, benzocaine, nitroprusside, isosorbide, or dapsone at screening
* History or clinical evidence of systolic heart failure, left ventricular dysfunction (LVEF <40%)
* Subjects reporting massive hemoptysis associated with the current illness or with radiologically proven pulmonary embolus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics
Locations (17):
- United States (17):
  - Banner University Medical Center, Phoenix, Arizona
  - Kaiser Permanente - Zion Medical Center, San Diego, California
  - Kaiser Permanente - San Diego Medical Center, San Diego, California
  - University of Miami Health System, Miami, Florida
  - The Lung Research Center (St. Luke's), Chesterfield, Missouri
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Houston Methodist, Houston, Texas
  - INOVA, Falls Church, Virginia
  - St. Francis Medical Center, Richmond, Virginia
  - Memorial Regional Medical Center, Richmond, Virginia
  - Chippenham Medical Center, Richmond, Virginia
  - Pulmonary Associates of Richmond, Richmond, Virginia
  - St. Mary's Hospital, Richmond, Virginia
  - Johnston-Willis Hospital, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Started | 95 | 96
Completed | 91 | 95
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo | Total
Number analyzed (Participants) | 95 | 96 | 191
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 age value missing in Placebo group
  Participants
    number analyzed (Participants) | 95 | 95 | 190
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 62 | 59 | 121
    >=65 years | 33 | 36 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (14.96) | 59.1 (13.72) | 58.6 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 44 | 92
  Male | 47 | 52 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 32 | 60
  Not Hispanic or Latino | 66 | 64 | 130
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 68 | 136
  Black or African American | 11 | 17 | 28
  Asian | 4 | 1 | 5
  America Indian or Alaska Native | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 95 | 96 | 191

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Died or Had Respiratory Failure
Description: The number of subjects who died or had respiratory failure through Day 28
Time Frame: Through Day 28
Population: All Randomized Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 95 | 96
Participants | 12 | 10
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide (iNO) vs Placebo; Test type: Superiority; p = 0.6316, Regression, Logistic; Odds Ratio (OR) = 0.36
Statistical Analysis 2: Comparison: Inhaled Nitric Oxide (iNO) vs Placebo; Test type: Superiority; p = 0.4127, Regression, Logistic — Odds ratio, 95% CI and p-value are from a logistic regression model modelling the response using the covariates treatment, age, number of co-morbidities and baseline oxygem level; Odds Ratio (OR) = 1.502, 95% CI 2-sided [0.567 to 3.977]

2. Secondary Outcome: Number of Subjects to Recover
Description: Number of subjects to recover, where recover is defined as attaining a NIAID Ordinal score of 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen or 8) Not hospitalized, no limitations on activities sustained through Day 28, or discharge from hospital without re admission for COVID.
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 95 | 96
Participants
  Recovered | 61 | 70
  Not Recovered | 34 | 26

3. Secondary Outcome: Clinical Status Using National Institute of Allergy and Infectious Diseases (NIAID) 8-point Ordinal Scale
Description: The assessment of clinical status at the first assessment of a study day. The scale is: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities.
Time Frame: Day 7
Population: All Randomized Analysis Set with NIAID scores at Day 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Pulsed Inhaled iNO 125 mcg/kg IBW/Hour: Pulsed inhaled iNO 125 mcg/kg IBW/hour INOpulse: Subjects will be treated by means of an INOpulse device using an INOpulse nasal cannula.
- Placebo N2, 99.999% Gas: Pulsed inhaled N2, 99.999% gas Placebo: Subjects will be treated by means of an INOpulse device using an INOpulse nasal cannula.
Arm/Group | Pulsed Inhaled iNO 125 mcg/kg IBW/Hour | Placebo N2, 99.999% Gas
Number analyzed (Participants) | 85 | 85
score on a scale | 5.28 (0.198) | 5.81 (0.192)

4. Secondary Outcome: Clinical Status Using National Institute of Allergy and Infectious Diseases (NIAID) 8-point Ordinal Scale
Description: as for outcome 3
Time Frame: Day 14
Population: All Randomized Analysis Set with NIAID scores at Day 14
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pulsed Inhaled iNO 125 mcg/kg IBW/Hour | Placebo N2, 99.999% Gas
Number analyzed (Participants) | 59 | 61
score on a scale | 6.22 (0.208) | 6.38 (0.202)

5. Secondary Outcome: Clinical Status Using National Institute of Allergy and Infectious Diseases (NIAID) 8-point Ordinal Scale
Description: as for outcome 3
Time Frame: Day 28
Population: All Randomized Analysis Set with NIAID scores at Day 28
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pulsed Inhaled iNO 125 mcg/kg IBW/Hour | Placebo N2, 99.999% Gas
Number analyzed (Participants) | 65 | 73
score on a scale | 6.56 (0.193) | 6.87 (0.186)

6. Secondary Outcome: Number of Subjects Discharged Alive From Hospital
Description: Number of subjects discharged alive from hospital through Day 28
Time Frame: Through Day 28
Population: (1) Discharged is defined as discharged alive from hospital through day 28. (2) For patients who were randomized but not treated, the date of randomization is used in place of the treatment start date.
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 95 | 96
Participants
  Discharged | 89 | 88
  Not Discharged | 6 | 7
  Missing Data | 0 | 1

7. Secondary Outcome: Duration of Hospitalization
Description: Duration of Hospitalization through Day 28
Time Frame: Through Day 28
Population: (1) Subject hospital duration will be defined as the time from Day 1 (start of study treatment) to the day of hospital discharge or Day 28 of treatment for patients who are still hospitalized. If a patient has expired on or before Day 27 of treatment, they will be assigned a value of 28 days. (2) For patients who were randomized but not treated, the date of randomization is used in place of the treatment start date.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 95 | 95
Days | 8.9 (6.58) | 8.1 (6.36)

8. Secondary Outcome: All Cause Mortality
Description: All cause mortality through Day 28
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 95 | 96
Participants | 5 | 1

9. Secondary Outcome: Difference in Proportion in RT-PCR Results at Discharge by Treatment Group
Description: Proportion of subjects with a positive RT-PCR result at baseline from a nasopharyngeal swab through Day 28 reported as a proportion of positive or negative RT-PCR testing.
Time Frame: Through Day 28
Population: Difference in converted RT-PCR Results at Discharge by Treatment Group. Only participants with a positive RT-PCR result at baseline are included in the analysis.
Measure: Number (95% Confidence Interval); unit: Proportion Converted
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 95 | 96
Proportion Converted
  Positive RT-PCR Result | 0.841 [0.751 to 0.932] | 0.812 [0.719 to 0.904]
  Negative RT-PCR Result | 0.159 [0.068 to 0.249] | 0.188 [0.096 to 0.281]
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide (iNO) vs Placebo; Test type: Superiority; p = 0.6635, Chi-squared

10. Other Pre Specified Outcome: Number of Subjects With Adverse Events Leading to Study Drug Discontinuation
Description: Number of subjects with adverse events leading to study drug discontinuation through Day 28
Time Frame: Through Day 28
Population: Full Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
Number analyzed (Participants) | 91 | 95
Participants | 11 | 11

ADVERSE EVENTS:
Time Frame: Collected during the study duration that includes 14 days within randomization to 30 days post last day of treatment (up to 28 days of blinded treatment)
Arm/Group | Inhaled Nitric Oxide (iNO) | Placebo
All-Cause Mortality (participants affected / at risk) | 5/91 | 1/95
Serious Adverse Events (participants affected / at risk) | 13/91 | 12/95
Other Adverse Events (participants affected / at risk) | 16/91 | 28/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (iNO) (N=91) | Placebo (N=95)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (iNO) (N=91) | Placebo (N=95)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Plural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum discolored (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
SARS-CoV-2 sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Renal and urinary disorders) | 0 (0) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Visual impariment (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 1 (1) | 1 (1)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT04421508/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT04421508/SAP_001.pdf